CLINICAL TRIAL: NCT00771329
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Dose, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of BIIB023 (Anti-TWEAK) Administered to Subjects With Rheumatoid Arthritis.
Brief Title: BIIB023 (Anti-TWEAK) in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Medical Director, Biogen Idec
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 211RA101
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2011-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — BIIB023

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): BIIB023
  Interventions: Drug: BIIB023
- 2 (Placebo Comparator)
  Interventions: Other: Placebo (sterile normal saline)

INTERVENTIONS:
Drug: BIIB023 — Single IV doses of BIIB023 in dose-escalating cohorts
  Other Names: Human glycosylated IgG1 monoclonal antibody
  Arms: 1
Other: Placebo (sterile normal saline) — Single IV dose of Placebo
  Arms: 2

SUMMARY:
Phase I study designed to determine the safety and tolerability of a single dose of BIIB023 administered intravenously versus placebo to subjects with RA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adult onset RA (functional class I-III) for at least 6 months
* Must have been treated with and be tolerating Methotrexate (5-25 mg/week) for 3 months, at a stable dose for at least 4 weeks
* Must have at least 4 swollen and tender joints due to rheumatoid arthritis

Exclusion Criteria:

* History of recurrent infections requiring antibiotic treatment within 12 months
* Serious local infection or systemic infection within 3 months
* Suffering from rheumatic or autoimmune disease other than RA
* History of cancer, heart failure, kidney disease, liver disease, HIV infection, tuberculosis or other serious illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Determine the safety and tolerability of single doses of BIIB023 administered intravenously (IV) to subjects with RA. | Baseline through Day 70

SECONDARY OUTCOMES:
• Estimate the pharmacokinetic (PK) parameters of single doses of BIIB023 administered IV to subjects with RA • Evaluate potential markers of pharmacodynamic (PD) action of BIIB023 and its biological effects | Day -1, 0 (at several timepoints), 1, 2, 7, 14, 21, 28, 42, 56 and Day 70

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - Research Site, Anniston, Alabama
  - Research Centre, Palm Desert, California
  - Research Site, Oklahoma City, Oklahoma
  - Research Centre, Duncansville, Pennsylvania
- Russia (2):
  - Research Centre, Moscow
  - Research Centre, Yaroslavl

REFERENCES:
- [Derived] Wisniacki N, Amaravadi L, Galluppi GR, Zheng TS, Zhang R, Kong J, Burkly LC. Safety, tolerability, pharmacokinetics, and pharmacodynamics of anti-TWEAK monoclonal antibody in patients with rheumatoid arthritis. Clin Ther. 2013 Aug;35(8):1137-49. doi: 10.1016/j.clinthera.2013.06.008. Epub 2013 Aug 6. PMID 23928094